CLINICAL TRIAL: NCT00671034
Title: A Pilot Study of Intravenous EZN-2285 (SC-PEG E. Coli L-asparaginase) or Intravenous Oncaspar® in the Treatment of Patients With High-Risk Acute Lymphoblastic Leukemia (ALL)
Brief Title: Calaspargase Pegol or Pegaspargase and Combination Chemotherapy in Treating Younger Patients With Newly Diagnosed High-Risk Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AALL07P4; NCI-2009-00317 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000594340; 08-606; COG-AALL07P4; AALL07P4 (Other: Children's Oncology Group); AALL07P4 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2008-05-01; First posted 2008-05-02 (Estimated); Results first posted 2018-09-06 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Acute Lymphoblastic Leukemia; Adult B Acute Lymphoblastic Leukemia; Childhood B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — calaspargase pegol; Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Mercaptopurine; azathiopurine; Methotrexate; merphos; pegaspargase; Prednisone; deltacortene; prednylidene; Radiotherapy; Radiation; Thioguanine; Vincristine

ARMS (2):
- Arm I (combination chemotherapy) (Experimental): Patients receive calaspargase pegol together with combination chemotherapy. Patients receive chemotherapy PO, IV, SC, and IT. Some patients also undergo radiation therapy to the head. Treatment may continue for up to 4 years.
  Interventions: Drug: Calaspargase Pegol-mknl; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Other: Pharmacological Study; Drug: Prednisone; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine Sulfate
- Arm II (combination chemotherapy) (Active Comparator): Patients receive pegaspargase together with combination chemotherapy. Patients receive chemotherapy PO, IV, SC, and IT. Some patients also undergo RT to the head. Treatment may continue for up to 4 years.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Pegaspargase; Other: Pharmacological Study; Drug: Prednisone; Radiation: Radiation Therapy; Drug: Thioguanine; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Calaspargase Pegol-mknl — Given IV
  Other Names: Asparaginase (Escherichia coli Isoenzyme II), Conjugate with alpha-(((2,5-Dioxo-1-pyrrolidinyl)oxy)carbonyl)-omega-methoxypoly(oxy-1,2-ethanediyl); Asparlas; Calaspargase Pegol; EZN-2285; SC-PEG E. Coli L-Asparaginase; Succinimidyl Carbonate Monomethoxypolyethylene Glycol E. coli L-Asparaginase
  Arms: Arm I (combination chemotherapy)
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IV, IT, PO, or SC
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Drug: Dexamethasone — Given PO or IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycadron; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decadron DP; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasone Intensol; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Dxevo; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; TaperDex; Visumetazone; ZoDex
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin HCl; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mercaptopurine — Given PO
  Other Names: 3H-Purine-6-thiol; 6 MP; 6 Thiohypoxanthine; 6 Thiopurine; 6-Mercaptopurine; 6-Mercaptopurine Monohydrate; 6-MP; 6-Purinethiol; 6-Thiopurine; 6-Thioxopurine; 6H-Purine-6-thione, 1,7-dihydro- (9CI); 7-Mercapto-1,3,4,6-tetrazaindene; Alti-Mercaptopurine; Azathiopurine; Bw 57-323H; Flocofil; Ismipur; Leukerin; Leupurin; Mercaleukim; Mercaleukin; Mercaptina; Mercaptopurinum; Mercapurin; Mern; NCI-C04886; Puri-Nethol; Purimethol; Purine, 6-mercapto-; Purine-6-thiol (8CI); Purine-6-thiol, monohydrate; Purinethiol; Purinethol; U-4748; WR-2785
Drug: Methotrexate — Given IV, IT, or PO
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Pegaspargase — Given IV
  Other Names: L-Asparaginase with Polyethylene Glycol; Oncaspar; Oncaspar-IV; PEG-Asparaginase; PEG-L-Asparaginase; PEG-L-Asparaginase (Enzon - Kyowa Hakko); PEGLA; Polyethylene Glycol L-Asparaginase; Polyethylene Glycol-L-Asparaginase
Other: Pharmacological Study — Correlative studies
Drug: Prednisone — Given IV or PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; Perrigo Prednisone; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisone Intensol; Prednisonum; Prednitone; Promifen; Rayos; Servisone; SK-Prednisone
Radiation: Radiation Therapy — Some patients undergo RT
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Thioguanine — Given PO
  Other Names: 2-Amino 6MP; 2-Amino-1,7-dihydro-6H-purine-6-thione; 2-Amino-6-mercaptopurine; 2-Amino-6-purinethiol; 2-Aminopurin-6-thiol; 2-Aminopurine-6(1H)-thione; 2-Aminopurine-6-thiol; 2-Aminopurine-6-thiol Hemihydrate; 2-Mercapto-6-aminopurine; 6-Amino-2-mercaptopurine; 6-Mercapto-2-aminopurine; 6-Mercaptoguanine; 6-TG; 6H-Purine-6-thione, 2-amino-1,7-dihydro- (9CI); BW 5071; Lanvis; Tabloid; Thioguanine Hemihydrate; Thioguanine Hydrate; Tioguanin; Tioguanine; Wellcome U3B; WR-1141; X 27
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine Sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate

SUMMARY:
This randomized clinical trial is studying giving calaspargase pegol together with combination chemotherapy to see how well it works compared with giving pegaspargase together with combination chemotherapy in treating younger patients with newly diagnosed high-risk acute lymphoblastic leukemia. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the pharmacokinetic comparability of EZN-2285 (calaspargase pegol) compared to Oncaspar (pegaspargase) given intravenously during induction and consolidation in patients with high-risk ALL receiving augmented Berlin-Frankfurt-Munster (BFM) therapy.

SECONDARY OBJECTIVES:

I. To describe the pharmacodynamics (PD) of EZN-2285 compared to Oncaspar given intravenously during induction and consolidation in patients with high-risk ALL receiving augmented BFM therapy.

II. To determine end of induction therapy day 29 minimal residual disease (MRD) for patients randomized to the EZN-2285 containing regimen compared to the Oncaspar® containing regimen.

III. To determine the complete remission (CR) rates for patients receiving EZN-2285 by day 29 of induction compared to Oncaspar.

IV. To assess event-free survival (EFS) associated with the administration of EZN-2285 given during augmented post Induction intensification therapy to patients with high-risk ALL compared to Oncaspar.

V. To determine the proportion of patients with an asparaginase level of at least 0.1 IU/mL and the proportion with at least 0.4 IU/mL on days 4, 15, 22 and 29 of induction compared to Oncaspar.

VI. To determine the plasma and cerebrospinal fluid (CSF) concentrations of asparagine after administration of EZN-2285 compared to Oncaspar.

VII. To assess the immunogenicity of EZN-2285 including the detection of binding and neutralizing antibodies compared to Oncaspar.

VIII. To assess the tolerability and toxicities associated with the administration of EZN-2285 given during augmented post induction intensification therapy to patients with high risk ALL compared to Oncaspar.

IX. To explore the relationship between the terminal pharmacokinetics (PK) of EZN-2285 and the presence of antibodies.

OUTLINE: This is a multicenter study. Patients are stratified according to response to induction therapy (slow early responders [SER] vs rapid early responders [RER]. Patients are randomized to 1 of 2 treatment arms in 2:1 ratio (arm I: arm II) (patients randomized to arm I receive study drug calaspargase pegol*; patients randomized to arm II receive study drug pegaspargase).

INDUCTION THERAPY** (ALL PATIENTS): Patients receive cytarabine intrathecally (IT) on day 1; vincristine intravenously (IV) and daunorubicin hydrochloride IV over 15 minutes on days 1, 8, 15, and 22; prednisone orally or IV twice daily (BID) on days 1-28; study drug IV over 1 hour on day 4; and methotrexate IT on days 8, 15*, 22*, and 29. Patients are assessed for response on day 8 and/or day 15 and day 29. Patients who achieve M1 marrow on day 8 or 15 and negative MRD (i.e., < 0.1%) on day 29 are considered RER. Patients who achieve M2 or M3 marrow on day 15 OR MRD >= 0.1% but < 1% on day 29 are considered SER. Patients with M3 bone marrow are removed from the study. RER and SER proceed to consolidation therapy. Patients with M2 marrow or M1 marrow with >= 1% MRD receive extended induction therapy. Patients also receive dexamethasone PO or IV BID on days 1-14 (patients < 10 years) or prednisone BID on days 1-28 (patients >= 10 years)

NOTE: *For patients with CNS3 disease only.

EXTENDED INDUCTION THERAPY**: Patients receive vincristine IV on days 1 and 8; prednisone orally (PO) or IV BID on days 1-14; daunorubicin hydrochloride IV over 15 minutes on day 1; and study drug IV over 1 hour on day 4. Patients are assessed for response on day 43. Patients who achieve M1 and MRD < 1% are treated as SER (proceed to consolidation therapy). All other patients are removed from study.

CONSOLIDATION THERAPY** (ALL PATIENTS): Beginning on day 36 (after completion of induction therapy) or after completion of extended induction therapy, patients (RER and SER) receive cyclophosphamide IV over 30 minutes on days 1 and 29; cytarabine IV or SC on days 1-4, 8-11, 29-32, and 36-39; mercaptopurine PO on days 1-14 and 29-42; vincristine IV on days 15, 22, 43, and 50; study drug IV over 1 hour on days 15 and 43; and methotrexate IT on days 1, 8, 15*, and 22*. Patients then proceed to interim maintenance I therapy.

NOTE: *Omit doses for patients with CNS3 disease.

INTERIM MAINTENANCE I** (ALL PATIENTS): Patients receive vincristine IV and methotrexate** IV on days 1, 11, 21, 31, and 41; study drug IV over 1 hour on days 2 and 22; and methotrexate IT on days 1 and 31. Patients then proceed to delayed intensification I therapy.

DELAYED INTENSIFICATION I** (ALL PATIENTS): Patients receive vincristine IV on days 1, 8, 15, 43, and 50; dexamethasone PO or IV BID on days 1-21 for patients age 1-9, or on days 1-7 and 15-21 for patients age >= 10; doxorubicin hydrochloride IV over 15 minutes on days 1, 8, and 15; study drug IV over 1 hour on days 4 and 43; cyclophosphamide IV over 30 minutes on day 29; cytarabine IV or subcutaneously (SC) on days 29-32 and 36-39; thioguanine PO on days 29-42; and methotrexate IT on days 1, 29, and 36. Patients treated as RER proceed to maintenance therapy. Patients treated as SER (i.e., patients with CNS3 disease at diagnosis, or pre-treated with steroids, or who are RERs with mixed lineage leukemia [MLL] gene rearrangements) proceed to interim maintenance II followed by delayed intensification II.

INTERIM MAINTENANCE II** (SER ONLY): Patients receive vincristine IV, methotrexate IV, study drug IV, and methotrexate IT as in interim maintenance I.

DELAYED INTENSIFICATION II** (SER ONLY): Beginning on day 29, patients (except patients with CNS3 disease) receive 8 daily fractions of cranial radiotherapy. All patients then receive vincristine IV, dexamethasone PO or IV, doxorubicin hydrochloride IV, study drug IV, cyclophosphamide IV, cytarabine IV or SC, thioguanine PO, and methotrexate IT as in delayed intensification I. Patients who were initially diagnosed with CNS3 disease receive cranial radiotherapy on days 1-5 and 8-12. Patients then proceed to maintenance therapy.

MAINTENANCE THERAPY** (ALL PATIENTS): Patients receive vincristine IV on days 1, 29, and 57; oral dexamethasone on days 1-5, 29-33, and 57-61; mercaptopurine PO on days 1-84; methotrexate IT on day 29; and methotrexate PO on days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78. Treatment repeats every 12 weeks for up to 2 years (for female patients) or up to 3 years (for male patients) from the start of interim maintenance I.

NOTE: ** As per amendment #4, most patients receive high-dose methotrexate instead of Capizzi methotrexate at most stages of therapy. CNS3 patients and SER patients who have received cranial irradiation receive planned therapy with no modifications.

NOTE: As per amendment #4, the maximum number of intrathecal treatments is limited by RER/SER/CNS3 status and gender.

Blood and cerebrospinal fluid samples are collected periodically for correlative studies, including immunogenicity, pharmacokinetic, and pharmacodynamic studies.

After completion of study therapy, patients are followed every 2 months for 2 years, every 3 months for 1 year, and then every 6-12 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be eligible for and enrolled on AALL08B1 or the successor classification study
* Patients must have newly diagnosed high-risk B lymphoblastic leukemia (World Health Organization [WHO] 2008 classification) (also termed B-precursor acute lymphoblastic leukemia)
* White blood cell (WBC) >= 50,000/μL for patients age 1-9 OR any WBC count for patients age 10-30 or for patients treated with prior steroids
* Patients shall have had no prior cytotoxic chemotherapy with the exception of steroids and intrathecal cytarabine; intrathecal chemotherapy with cytarabine is allowed prior to registration for patient convenience; this is usually done at the time of the diagnostic bone marrow or venous line placement to avoid a second lumbar puncture; (Note: the CNS status must be determined based on a sample obtained prior to administration of any systemic or intrathecal chemotherapy, except for steroid pretreatment) systemic chemotherapy must begin within 72 hours of this intrathecal therapy
* Patients receiving prior steroid therapy are eligible for this study; the dose and duration of previous steroid therapy should be carefully documented
* Pregnancy tests with a negative result must be obtained in all post-menarchal females
* Lactating females must agree that they will not breastfeed a child while on this study

Exclusion Criteria:

* Patients with Down syndrome are excluded from this study
* Patients with testicular leukemia at diagnosis are excluded from this study
* Pregnant female patients are excluded from this study

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 166 (Actual)
Dates: Start 2008-07-21 (Actual); Primary Completion 2011-02-01 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne L Angiolillo, Principal Investigator — Children's Oncology Group
Locations (27):
- United States (27):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Connecticut, Farmington, Connecticut
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] Schore RJ, Devidas M, Bleyer A, Reaman GH, Winick N, Loh ML, Raetz EA, Carroll WL, Hunger SP, Angiolillo AL. Plasma asparaginase activity and asparagine depletion in acute lymphoblastic leukemia patients treated with pegaspargase on Children's Oncology Group AALL07P4. Leuk Lymphoma. 2019 Jul;60(7):1740-1748. doi: 10.1080/10428194.2018.1542146. Epub 2019 Jan 10. PMID 30626253

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Calaspargase Pegol 2100); Arm II (Calaspargase Pegol 2500): Patients receive calaspargase pegol together with combination chemotherapy. Patients receive chemotherapy PO, IV, SC, and IT. Some patients also undergo radiation therapy to the head. Treatment may continue for up to 3 1/2 years.
- Arm III (Pegaspargase 2500): Patients receive pegaspargase together with combination chemotherapy. Patients receive chemotherapy PO, IV, SC, and IT. Some patients also undergo RT to the head. Treatment may continue for up to 3 1/2 years.
Period: Overall Study
Arm/Group | Arm I (Calaspargase Pegol 2100) | Arm II (Calaspargase Pegol 2500) | Arm III (Pegaspargase 2500)
Started | 69 | 42 | 55
Completed | 30 | 22 | 31
Not Completed | 39 | 20 | 24
Not completed — Adverse Event | 5 | 7 | 1
Not completed — Death | 3 | 2 | 1
Not completed — Physician Decision | 12 | 4 | 5
Not completed — VHR ALL feature | 8 | 3 | 5
Not completed — Refusal | 5 | 3 | 5
Not completed — includes Alternative therapy, etc. | 6 | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Arm I (Calaspargase Pegol 2100): calaspargase pegol 2100
- Arm II (Calaspargase Pegol 2500): calaspargase pegol 2500
- Arm III (Pegaspargase 2500): pegaspargase 2500
- Total: Total of all reporting groups
Arm/Group | Arm I (Calaspargase Pegol 2100) | Arm II (Calaspargase Pegol 2500) | Arm III (Pegaspargase 2500) | Total
Number analyzed (Participants) | 69 | 42 | 55 | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 62 | 40 | 51 | 153
  Between 18 and 65 years | 7 | 2 | 4 | 13
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.9 (5.58) | 9.9 (6.09) | 10.79 (5.54) | 11.3 (5.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 28 | 23 | 82
  Male | 38 | 14 | 32 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 12 | 18 | 44
  Not Hispanic or Latino | 53 | 28 | 35 | 116
  Unknown or Not Reported | 2 | 2 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 4 | 1 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 4 | 1 | 6 | 11
  White | 56 | 35 | 43 | 134
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK) (Half-life of SC-PEG E. Coli L-asparaginase (EZN-2285) Compared to Pegaspargase During Induction and Consolidation Therapy)
Description: Mean half-life of plasma asparaginase during consolidation and Induction; half-life is defined as the time taken for drug concentration to decrease by half.
Time Frame: Post Day 29 of Induction and Post Day 22 of Consolidation
Population: Analysis restricted to patients who had PK data collected
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Arm II ( Calaspargase Pegol 2500): Patients receive calaspargase pegol together with combination chemotherapy. Patients receive chemotherapy PO, IV, SC, and IT. Some patients also undergo radiation therapy to the head. Treatment may continue for up to 3 1/2 years.
Arm/Group | Arm I (Calaspargase Pegol 2100) | Arm II ( Calaspargase Pegol 2500) | Arm III (Pegaspargase 2500)
Number analyzed (Participants) | 69 | 42 | 54
hours
  Asparaginase half-life during Consolidation: number analyzed (Participants) | 24 | 17 | 24
  Asparaginase half-life during Consolidation | 415.8 (148.51) | 355.9 (133.0) | 117.2 (49.36)
  Asparaginase half-life during Induction: number analyzed (Participants) | 58 | 40 | 43
  Asparaginase half-life during Induction | 305.1 (98.33) | 321.5 (118.22) | 126.9 (50.51)

2. Secondary Outcome: Pharmacodynamics (PD)
Description: Plasma Asparaginase Concentration During consolidation and induction.
Time Frame: Day 29 of consolidation and induction
Population: Patients who had data collected
Measure: Median (Standard Deviation); unit: mIU/mL
Arm/Group | Arm I (Calaspargase Pegol 2100) | Arm II (Calaspargase Pegol 2500) | Arm III (Pegaspargase 2500)
Number analyzed (Participants) | 69 | 42 | 54
mIU/mL
  Plasma Asparaginase Concentration- Consolidation: number analyzed (Participants) | 33 | 18 | 30
  Plasma Asparaginase Concentration- Consolidation | 575.9 (233.91) | 617.2 (321.41) | 562.1 (296.82)
  Plasma Asparaginase Concentration- Induction: number analyzed (Participants) | 59 | 40 | 42
  Plasma Asparaginase Concentration- Induction | 271.6 (118.17) | 339.6 (126.83) | 72.8 (47.94)

3. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD)<0.01% at the End of Induction
Description: Percentage of participants with Negative MRD (MRD<0.01%).
Time Frame: End of induction (Day 29)
Population: Patients who had data collected.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm I (Calaspargase Pegol 2100) | Arm II (Calaspargase Pegol 2500) | Arm III (Pegaspargase 2500)
Number analyzed (Participants) | 62 | 40 | 47
Percentage of participants | 65.2 [52.4 to 76.5] | 81 [65.9 to 91.4] | 72.5 [58.3 to 84.1]

4. Secondary Outcome: Percentage of Participants With Complete Remission at the End of Induction
Description: Complete Remission (CR) rate; where CR is defined as M1 marrow (< 5% lymphoblasts in the bone marrow)
Time Frame: End of induction (Day 29)
Population: Patients who had data collected
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm I (Calaspargase Pegol 2100) | Arm II (Calaspargase Pegol 2500) | Arm III (Pegaspargase 2500)
Number analyzed (Participants) | 66 | 42 | 51
Percentage of participants | 92.4 [83.2 to 97.5] | 97.6 [87.4 to 99.9] | 94.1 [83.8 to 98.8]

5. Secondary Outcome: Percentage of Participants With Event-free Survival (EFS)
Description: Percentage of participants who were event free. Event Free Probability defined as time from randomization at study entry to first event (induction failure, induction death, relapse, second malignant neoplasm, remission death) or date of last contact for subjects who are event-free.
Time Frame: 5 Years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm I (Calaspargase Pegol 2100) | Arm II (Calaspargase Pegol 2500) | Arm III (Pegaspargase 2500)
Number analyzed (Participants) | 69 | 42 | 54
Percentage of participants | 72.35 [60.98 to 83.72] | 80.8 [68.3 to 93.3] | 79.34 [67.56 to 91.12]

6. Secondary Outcome: Asparaginase Level
Description: The proportion of patients with an asparaginase level of at least 0.1 IU/mL and the proportion with at least 0.4 IU/mL on Days 4, 15, 22 and 29 of Induction compared to Oncaspar
Time Frame: Days 4, 15, 22 and 29 of Induction
Population: Patients who had data collected.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm I (Calaspargase Pegol 2100) | Arm II (Calaspargase Pegol 2500) | Arm III (Pegaspargase 2500)
Number analyzed (Participants) | 69 | 42 | 54
percentage of patients
  Level at least 0.1 IU/mL day 4: number analyzed (Participants) | 62 | 40 | 43
  Level at least 0.1 IU/mL day 4 | 0 [0.0 to 8.2] | 0 [0.0 to 8.8] | 0 [0.0 to 5.8]
  Level at least 0.1 IU/mL day 15: number analyzed (Participants) | 62 | 40 | 43
  Level at least 0.1 IU/mL day 15 | 98.4 [91.3 to 100.0] | 100 [91.2 to 100] | 100 [98.1 to 100]
  Level at least 0.1 IU/mL day 22: number analyzed (Participants) | 56 | 40 | 41
  Level at least 0.1 IU/mL day 22 | 98.2 [78.1 to 98.5] | 100 [91.2 to 100] | 95.1 [77.9 to 97.4]
  Level at least 0.1 IU/mL day 29: number analyzed (Participants) | 59 | 40 | 42
  Level at least 0.1 IU/mL day 29 | 94.9 [80.1 to 96.4] | 95.0 [83.1 to 99.4] | 28.6 [15.3 to 43.7]
  Level at least 0.4 IU/mL day 4: number analyzed (Participants) | 62 | 40 | 43
  Level at least 0.4 IU/mL day 4 | 0 [0.0 to 8.2] | 0 [0.0 to 8.8] | 0 [0.0 to 5.8]
  Level at least 0.4 IU/mL day 15: number analyzed (Participants) | 62 | 40 | 43
  Level at least 0.4 IU/mL day 15 | 75.8 [63.3 to 85.8] | 95.0 [83.1 to 99.4] | 93.0 [80.9 to 98.5]
  Level at least 0.4 IU/mL day 22: number analyzed (Participants) | 56 | 40 | 41
  Level at least 0.4 IU/mL day 22 | 37.5 [22.3 to 47.0] | 62.5 [45.8 to 77.3] | 14.6 [5.3 to 27.9]
  Level at least 0.4 IU/mL day 29: number analyzed (Participants) | 59 | 40 | 42
  Level at least 0.4 IU/mL day 29 | 13.6 [5.7 to 23.9] | 27.5 [14.6 to 43.9] | 0 [0.0 to 8.2]

7. Secondary Outcome: Plasma and CSF Concentrations of Asparagine in ug/ml
Description: The plasma and CSF concentrations of asparagine in ug/ml after administration of EZN-2285 compared to Oncaspar.
Time Frame: 25 Days Post-dose (Day 29)
Population: Patients who had data collected.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Arm I (Calaspargase Pegol 2100) | Arm II (Calaspargase Pegol 2500) | Arm III (Pegaspargase 2500)
Number analyzed (Participants) | 69 | 42 | 54
ug/mL
  CSF asparagine concentration (ug/mL): number analyzed (Participants) | 51 | 38 | 38
  CSF asparagine concentration (ug/mL) | 0.2 (0.108) | 0.19 (0.086) | 0.26 (0.26)
  Plasma asparagine concentration (ug/mL): number analyzed (Participants) | 55 | 39 | 41
  Plasma asparagine concentration (ug/mL) | 0.2 (0.784) | 0.25 (1.231) | 0.83 (2.195)

8. Secondary Outcome: Immunogenicity
Description: Number of Patients with Positive Immunogenicity tests
Time Frame: 25 Days Post-dose (Day 29)
Population: Patients who had data collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Calaspargase Pegol 2100) | Arm II (Calaspargase Pegol 2500) | Arm III (Pegaspargase 2500)
Number analyzed (Participants) | 69 | 42 | 54
Participants | 2 | 2 | 4

9. Secondary Outcome: Toxicities During Post Induction Intensification Therapy (All Grades)
Description: The calculation of AE incidence will be based on the number of patients per AE category. For each patient who has multiple AEs classified to the same category, that patient will be tabulated under the worst toxicity grade for that AE category. The incidence of AEs will be tabulated by treatment arm and by organ class. Special attention will be paid to hypersensitivity, pancreatitis, coagulopathy, infection, neurologic dysfunction and thromboembolic events.
Time Frame: Up to 5 years
Population: Patients who had data collected. International normalized ratio (INR). Activated partial thromboplastin (APT)
Measure: Number; unit: Percentage of participants
Arm/Group | Arm I (Calaspargase Pegol 2100) | Arm II (Calaspargase Pegol 2500) | Arm III (Pegaspargase 2500)
Number analyzed (Participants) | 49 | 33 | 43
Percentage of participants
  Alergic Reaction - Consolidation | 20.4 | 27.3 | 23.3
  Alergic Reaction - Delayed Intensification I: number analyzed (Participants) | 45 | 26 | 38
  Alergic Reaction - Delayed Intensification I | 4.4 | 0.0 | 0.0
  Alergic Reaction - Interim Maintenance I: number analyzed (Participants) | 46 | 29 | 39
  Alergic Reaction - Interim Maintenance I | 0.0 | 0.0 | 2.1
  CNS - Consolidation | 0.0 | 0.0 | 0.0
  CNS - Delayed Intensification I: number analyzed (Participants) | 45 | 26 | 38
  CNS - Delayed Intensification I | 0.0 | 3.8 | 2.6
  CNS - Interim Maintenance I: number analyzed (Participants) | 46 | 29 | 39
  CNS - Interim Maintenance I | 0.0 | 0.0 | 0.0
  Hyperbilirubinemia - Consolidation | 53.1 | 45.5 | 30.2
  Hyperbilirubinemia - Delayed Intensification I: number analyzed (Participants) | 45 | 26 | 38
  Hyperbilirubinemia - Delayed Intensification I | 28.9 | 38.5 | 10.5
  Hyperbilirubinemia - Interim Maintenance I: number analyzed (Participants) | 46 | 29 | 39
  Hyperbilirubinemia - Interim Maintenance I | 41.3 | 27.6 | 33.3
  Hyperglycemia - Consolidation | 44.9 | 42.4 | 46.5
  Hyperglycemia - Delayed Intensification I: number analyzed (Participants) | 45 | 26 | 38
  Hyperglycemia - Delayed Intensification I | 44.4 | 61.5 | 36.8
  Hyperglycemia - Interim Maintenance I: number analyzed (Participants) | 46 | 29 | 39
  Hyperglycemia - Interim Maintenance I | 34.8 | 44.8 | 33.3
  Hyperlipidemia - Consolidation | 2.0 | 3.0 | 7.0
  Hyperlipidemia - Delayed Intensification I: number analyzed (Participants) | 45 | 26 | 38
  Hyperlipidemia - Delayed Intensification I | 2.2 | 0.0 | 0.0
  Hyperlipidemia - Interim Maintenance I: number analyzed (Participants) | 46 | 29 | 39
  Hyperlipidemia - Interim Maintenance I | 2.2 | 3.4 | 2.6
  % patients w/INR increase - Consolidation | 6.1 | 3.0 | 7.0
  % pts w/INR increase - Delayed Intensification I: number analyzed (Participants) | 45 | 26 | 38
  % pts w/INR increase - Delayed Intensification I | 6.7 | 3.8 | 0.0
  % patients w/INR increase - Interim Maintenance I: number analyzed (Participants) | 46 | 29 | 39
  % patients w/INR increase - Interim Maintenance I | 2.2 | 0.0 | 2.6
  Pancreatitis - Consolidation | 10.2 | 6.1 | 7.0
  Pancreatitis -Delayed Intensification I: number analyzed (Participants) | 45 | 26 | 38
  Pancreatitis -Delayed Intensification I | 2.2 | 7.7 | 0.0
  Pancreatitis - Interim Maintenance I: number analyzed (Participants) | 46 | 29 | 39
  Pancreatitis - Interim Maintenance I | 2.2 | 3.4 | 2.6
  % pts w/prolongation of APT time - Consolidation | 8.2 | 9.1 | 7.0
  % pts w/prolongation APT time -Delayed Intension I: number analyzed (Participants) | 45 | 26 | 38
  % pts w/prolongation APT time -Delayed Intension I | 8.9 | 26.9 | 18.4
  %pts w/prolongation APT time-Interim maintenance I: number analyzed (Participants) | 46 | 29 | 39
  %pts w/prolongation APT time-Interim maintenance I | 6.5 | 6.9 | 7.7
  Thrombosis - Consolidation | 0.0 | 0.0 | 2.3
  Thrombosis - Delayed Intensification I: number analyzed (Participants) | 45 | 26 | 38
  Thrombosis - Delayed Intensification I | 2.2 | 0.0 | 0.0
  Thrombosis - Interim Maintenance I: number analyzed (Participants) | 46 | 29 | 39
  Thrombosis - Interim Maintenance I | 0.0 | 0.0 | 0.0

10. Secondary Outcome: Relationship Between PK and Presence of Antibodies
Description: Patients with presence of Antibodies.
Time Frame: Day 29 of consolidation
Population: These data will never be collected.
Arm/Group | Arm I (Calaspargase Pegol 2100) | Arm II (Calaspargase Pegol 2500) | Arm III (Pegaspargase 2500)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I (Calaspargase Pegol 2100) | Arm II (Calaspargase Pegol 2500) | Arm III (Pegaspargase 2500)
Serious Adverse Events (participants affected / at risk) | 54/69 | 34/42 | 32/54
Other Adverse Events (participants affected / at risk) | 64/69 | 40/42 | 51/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Calaspargase Pegol 2100) (N=69) | Arm II (Calaspargase Pegol 2500) (N=42) | Arm III (Pegaspargase 2500) (N=54)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 11 (14) | 7 (7) | 4 (4)
Anal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 3 (5) | 0 (0) | 1 (1)
Pancreatic necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 8 (8) | 6 (6) | 4 (4)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Death NOS (General disorders) | 4 (4) | 1 (1) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0) | 1 (1)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 2 (2) | 1 (2)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylaxis (Immune system disorders) | 13 (13) | 11 (11) | 10 (11)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 14 (17) | 8 (10) | 4 (6)
Infective myositis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3) | 3 (3) | 3 (3)
Alanine aminotransferase increased (Investigations) | 4 (4) | 2 (3) | 5 (6)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 2 (2) | 4 (4)
Blood bilirubin increased (Investigations) | 12 (13) | 8 (10) | 10 (12)
CPK increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 2 (4) | 2 (4) | 3 (5)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Fibrinogen decreased (Investigations) | 4 (4) | 3 (3) | 3 (3)
GGT increased (Investigations) | 1 (1) | 2 (2) | 1 (1)
INR increased (Investigations) | 1 (1) | 3 (3) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 7 (7) | 4 (4) | 4 (4)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (2) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 6 (6) | 1 (1) | 1 (2)
Serum amylase increased (Investigations) | 8 (8) | 1 (1) | 2 (2)
Weight loss (Investigations) | 3 (3) | 2 (2) | 1 (7)
White blood cell decreased (Investigations) | 1 (1) | 2 (2) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 5 (7) | 1 (10) | 1 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 3 (4)
Glucose intolerance (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 21 (27) | 14 (16) | 12 (17)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 (7) | 4 (7) | 6 (10)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (6) | 2 (2) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Arachnoiditis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 2 (2) | 1 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 2 (2) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 2 (2) | 3 (3)
Agitation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 7 (7) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 5 (7) | 0 (0) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Calaspargase Pegol 2100) (N=69) | Arm II (Calaspargase Pegol 2500) (N=42) | Arm III (Pegaspargase 2500) (N=54)
Anemia (Blood and lymphatic system disorders) | 18 (23) | 16 (27) | 23 (33)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 37 (88) | 26 (60) | 31 (56)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 1 (2) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 8 (8) | 6 (9)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (10) | 4 (6) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 16 (23) | 4 (5) | 7 (9)
Nausea (Gastrointestinal disorders) | 9 (10) | 3 (3) | 2 (3)
Oral hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 6 (7) | 1 (1) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (7) | 2 (3) | 5 (5)
Facial pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (4) | 3 (4) | 2 (2)
Fever (General disorders) | 3 (4) | 5 (5) | 3 (3)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 3 (3) | 2 (2)
Pain (General disorders) | 5 (10) | 1 (1) | 2 (3)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylaxis (Immune system disorders) | 2 (2) | 2 (2) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 5 (6) | 1 (1) | 1 (2)
Infections and infestations - Other, specify (Infections and infestations) | 30 (57) | 23 (55) | 18 (39)
Infective myositis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 8 (9) | 3 (3) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Pancreas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 3 (4) | 2 (2) | 2 (3)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (5) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 25 (71) | 22 (47) | 27 (73)
Alkaline phosphatase increased (Investigations) | 3 (3) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 10 (19) | 11 (15) | 14 (30)
Blood bilirubin increased (Investigations) | 8 (8) | 3 (3) | 3 (3)
Cholesterol high (Investigations) | 0 (0) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 0 (0) | 1 (1)
GGT increased (Investigations) | 3 (3) | 3 (7) | 7 (19)
Investigations - Other, specify (Investigations) | 1 (1) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 2 (2) | 7 (8) | 5 (5)
Lymphocyte count decreased (Investigations) | 0 (0) | 4 (4) | 0 (0)
Neutrophil count decreased (Investigations) | 44 (121) | 29 (82) | 36 (92)
Platelet count decreased (Investigations) | 30 (52) | 20 (37) | 22 (33)
Serum amylase increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Weight gain (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight loss (Investigations) | 5 (5) | 4 (5) | 1 (1)
White blood cell decreased (Investigations) | 19 (27) | 16 (34) | 18 (45)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (3)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 11 (13) | 8 (11) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 3 (5)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 18 (36) | 11 (12) | 9 (18)
Hyperkalemia (Metabolism and nutrition disorders) | 9 (10) | 2 (3) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (11) | 8 (9) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 13 (18) | 4 (4) | 11 (15)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 25 (40) | 15 (18) | 14 (21)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 12 (12) | 8 (10) | 8 (10)
Hypophosphatemia (Metabolism and nutrition disorders) | 9 (10) | 2 (2) | 3 (3)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (7)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 2 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 4 (4)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (5) | 4 (5) | 3 (3)
Abducens nerve disorder (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (3)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 7 (8) | 7 (7)
Hypoglossal nerve disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vagus nerve disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vasovagal reaction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (2) | 0 (0) | 2 (2)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Uterine hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (10) | 3 (3) | 5 (5)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 4 (4) | 4 (5) | 3 (3)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Data is not and never will be available for Outcome Measure 10, Relationship between PK and presence of antibodies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain sponsor approval.